CLINICAL TRIAL: NCT01668485
Title: Metabolic Studies in Type 1 Diabetic Patients After Allogenic Intraportal Islet Transplantation.
Brief Title: Mechanisms of Glucose Counterregulation in Pancreatic Islet Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Thomas Linn, Professor Dr. med., University of Giessen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: T1DM/ITX
Record Dates: First submitted 2012-08-13; First posted 2012-08-20 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; hypoglycemia counterregulation,; pancreatic islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Islet transplant recipients (Experimental): Hypoglycemic and euglycemic glucose clamp
  Interventions: Procedure: Hypoglycemic and euglycemic glucose clamp
- Type 1 diabetic subjects (Placebo Comparator): Hypoglycemic and euglycemic glucose clamp.
  Interventions: Procedure: Hypoglycemic and euglycemic glucose clamp
- Non-diabetic subjects (Active Comparator): Hypoglycemic and euglycemic glucose clamp
  Interventions: Procedure: Hypoglycemic and euglycemic glucose clamp

INTERVENTIONS:
Procedure: Hypoglycemic and euglycemic glucose clamp — Each study participant will be subjected to a continuous infusion of insulin at a rate of 0.8 mU·kg-1·min-1 to induce hypoglycemia (blood glucose 2.8-3 mmol/l) for 30 minutes. At least two weeks later an identical insulin infusion will be administered and euglycemia (blood glucose 5 mmol/l) will be targeted. The order of these interventions will be subject to randomization.

SUMMARY:
Pancreatic islet transplantation improves glucose counterregulation and stabilizes glycemic control in patients with type 1 diabetes mellitus prone to severe hypoglycemia even if insulin independence is not achieved. However, the extent and underlying metabolic pathways of this improvement are unknown. Investigators therefore compare systemic glucose turnover including lactate gluconeogenesis and muscle glucose utilization, between insulin-requiring islet transplant recipients, matched type 1 diabetic subjects who did not receive islet transplantation, and matched healthy non-diabetic subjects.

DETAILED DESCRIPTION:
Subjects (n=12 each group) undergo a hypoglycemic and a euglycemic hyperinsulinemic clamp in a randomized fashion. Systemic and skeletal muscle glucose and lactate kinetics are assessed using a combination of isotopic and forearm balance techniques.

ELIGIBILITY:
T1DM/ITX+

Inclusion Criteria:

* Type 1 Diabetes
* Pancreatic islet transplantation

Exclusion Criteria:

* Type 2 Diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-11; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Whole body glucose counterregulation | 6-8 weeks
  Whole body glucose counterregulation is the difference in glucose infusion rates required to maintain the glycemic goal between the hypoglycemic and euglycemic clamp. Clamps were performed at two time points at least two weeks apart. Participants will be followed for the duration of 6-8 weeks to perform the hypoglycemic and euglycemic clamp tests.

SECONDARY OUTCOMES:
Systemic glucose release | 6-8 weeks
  Systemic glucose release is the amount of glucose released primarily from the liver into the blood compartment during a given time. The unit of measure is μmol/kg/min.
  Participants will be followed for the duration of 6-8 weeks to perform the hypoglycemic and euglycemic clamp tests that will yield this parameter.
Skeletal muscle glucose disposal | 6-8 weeks
  Participants will be followed for the duration of 6-8 weeks to perform the euglycemic and hypoglycemic clamp tests. The unit of measure of this parameters is μmol/kg/min.
Gluconeogenesis from lactate | 6-8 weeks
  This parameter is determined by labelled lactate infused into the proband. The rate of the de novo synthesis of glucose (gluconeogenesis) is determined by the degree of incorporation of the lactate label into glucose molecules. The unit of measure of this parameter is μmol/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Linn, MD, Principal Investigator — Justus Liebig University
Locations (1):
- Justus Liebig University, Giessen, Hessia, Germany

REFERENCES:
- [Derived] Ang M, Meyer C, Brendel MD, Bretzel RG, Linn T. Magnitude and mechanisms of glucose counterregulation following islet transplantation in patients with type 1 diabetes suffering from severe hypoglycaemic episodes. Diabetologia. 2014 Mar;57(3):623-32. doi: 10.1007/s00125-013-3120-9. Epub 2013 Dec 5. PMID 24305963